CLINICAL TRIAL: NCT06323070
Title: Effects of Watermelon or Low-fat Cookie Consumption on Wellness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS-2023-0281
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-fat cookies (Active Comparator): Subjects consume 100 kcal of low-fat cookies daily for 4 weeks.
  Interventions: Other: Low-fat cookies
- Watermelon (Experimental): Subjects consume 100 kcal of watermelon daily for 4 weeks.
  Interventions: Other: Watermelon

INTERVENTIONS:
Other: Low-fat cookies — To determine the effects of low-fat cookie consumption on physiological indicators of wellness regarding sexual, skin, and gut health
  Arms: Low-fat cookies
Other: Watermelon — To determine the effects of watermelon consumption on physiological indicators of wellness regarding sexual, skin, and gut health
  Arms: Watermelon

SUMMARY:
The objective of the proposed research is to determine the effects of fresh watermelon consumption on physiological indicators of wellness regarding sexual, skin and gut health in adults.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects
* BMI 20-40 kg/m2

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required antibiotics use
* Required dietary supplement use
* Required medication of metabolic disorders, mental health and sexual health
* Allergy to watermelon or wheat

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of sexual health questionnaire scores | Baseline and week 4
  Change of sexual health questionnaire scores will be determined to examine effects of watermelon consumption vs low-fat cookies.
Change of skin hydration scores | Baseline, 1 min post application and week 4 consumption
  Change of skin hydration scores will be determined to examine effects of watermelon consumption vs low-fat cookies.
Change of microbiome diversity | Baseline and week 4
  Change of skin hydration scores will be determined to examine effects of watermelon consumption vs low-fat cookies.

SECONDARY OUTCOMES:
Change of depression questionnaire scores | Baseline and week 4
  Change of depression questionnaire scores will be determined to examine effects of watermelon consumption vs low-fat cookies.

CONTACTS AND LOCATIONS:
Overall Officials: Mee Young Hong, PhD, Principal Investigator — San Diego State University
Locations (1):
- School of Exercise and Nutritional Sciences, San Diego, California, United States